CLINICAL TRIAL: NCT04731090
Title: Effect of Standard Antibiotic Prophylaxis Versus Enhanced Prophylactic Measures on Rate of Urinary Tract Infection After Flexible Ureteroscopy
Brief Title: Standard Antibiotic Versus Enhanced Prophylactic Measures on Rate of Urinary Tract Infection After Flexible Ureteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N2113
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections | interventions — Fluoroquinolones; Anti-Bacterial Agents; Antibiotic Prophylaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard antibiotic prophylaxis (Active Comparator): IV fluoroquinolone 1 hour preoperatively and oral antibiotics were used for 24h postoperatively.
  Interventions: Drug: IV fluoroquinolone 1 hour preoperatively and oral antibiotics for 24h postoperatively.
- enhanced prophylaxis (Experimental): Patients had urine culture 10 days before the procedure. In addition to the antibiotic prophylaxis, hydrophilic-coated ureteral access sheaths were systematically used.
  Interventions: Other: Urine culture, antibiotic prophylaxis and hydrophilic-coated ureteral access sheaths

INTERVENTIONS:
Drug: IV fluoroquinolone 1 hour preoperatively and oral antibiotics for 24h postoperatively. — IV fluoroquinolone 1 hour preoperatively and oral antibiotics for 24h postoperatively.
  Arms: Standard antibiotic prophylaxis
Other: Urine culture, antibiotic prophylaxis and hydrophilic-coated ureteral access sheaths — Patients had urine culture 10 days before the procedure. In addition to the antibiotic prophylaxis, hydrophilic-coated ureteral access sheaths were systematically used.
  Arms: enhanced prophylaxis

SUMMARY:
Background and aim: Urinary tract infections (UTIs) are commonly seen after flexible ureteroscopy. Prevention of UTIs remains controversial. The present randomized study aimed to compare the rate of post-procedural UTI in patients subjected to the standard antibiotic prophylaxis alone versus enhanced prophylactic measures.

Patients and methods: The study included 100 patients subjected to fURS for management of ureteral and/or renal stones. Patients were equally and randomly allocated into one of the two treatment groups using randomly computer-generated allocation tables and concealed envelope technique. Treatment groups included standard antibiotic prophylaxis group and enhanced prophylaxis group. Patients in the standard antibiotic prophylaxis group IV fluoroquinolone 1 hour preoperatively and oral antibiotics were used for 24h postoperatively. In the enhanced prophylaxis group, patients had urine culture 10 days before the procedure. In addition to the antibiotic prophylaxis, hydrophilic-coated ureteral access sheaths were systematically used.

ELIGIBILITY:
Inclusion Criteria:

* All patients subjected to flexible ureteroscopy for management of ureteral and/or renal stones.

Exclusion Criteria:

* Symptomatic urinary tract infection.
* Use of rigid ureteroscopy and antegrade ureteroscopy.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Urinary tract infection | 30-day postoperative
  Postoperative UTI was defined as the occurrence of a temperature higher than 38 °C associated with pyuria and/or bacteriuria without any other focal infectious sites.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elhelaly, Principal Investigator — Al-Azhar Universiy
Locations (1):
- Armed forced Hospital, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No